CLINICAL TRIAL: NCT01187615
Title: An Open-label, Multi-center, Non-randomized Phase Ib Study to Investigate the Safety, Efficacy, and Pharmacokinetics of BAY 73-4506 "Regorafenib", Administered in Combination With Pemetrexed and Cisplatin in Patients With Advanced Nonsquamous Non-Small Cell Lung Cancer
Brief Title: Determination of Safety, Efficacy, and Pharmacokinetics of "Regorafenib" Combined With Pemetrexed and Cisplatin in Patients With Nonsquamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14458
Record Dates: First submitted 2010-07-16; First posted 2010-08-24 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Nonsquamous Non-small cell lung cancer; Phase I
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — regorafenib; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506) - sequential / Cisplatin / Pemetrexed
- Arm 2 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506) - continuous / Cisplatin / Pemetrexed

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) - sequential / Cisplatin / Pemetrexed — In Part A of this trial, regorafenib will be administered in a sequential dosing with a seven day wash out period before the next infusion of pemetrexed and cisplatin. Regorafenib will be administered at a dose of 160 mg qd from Day 2 to Day 14 followed by a 7 days break. Pharmacokinetics of regorafenib will be assessed on Day 14 of Cycle 1 and Day 1 of Cycle 2.
  Arms: Arm 1
Drug: Regorafenib (BAY73-4506) - continuous / Cisplatin / Pemetrexed — In Part B of this trial, regorafenib will be administered continuously from Day 1 to Day 21. Only in Cycle 1, regorafenib dosing will start on Day 2 in order to assess the pharmacokinetics of pemetrexed and cisplatin without concomitant regorafenib dosing. Pharmacokinetics of regorafenib will be assessed on Day 21 of Cycle 1 and on Day 1 of Cycle 2.
  Arms: Arm 2

SUMMARY:
This is a multi-center, open-label, non-randomized Phase I study to define the safety profile, maximum tolerated dose (MTD) and potential pharmacokinetic interaction of regorafenib in combination with pemetrexed and cisplatin in patients with Stage IIIB or Stage IV nonsquamous Non-Small Cell Lung Cancer (NSCLC) and to determine the impact of the combined administration on the pharmacokinetics of regorafenib, pemetrexed, and cisplatin.

In Part A of this trial, regorafenib will be administered in a sequential dosing with a seven day wash out period before the next infusion of pemetrexed and cisplatin. Regorafenib will be administered at a dose of 160 mg qd from Day 2 to Day 14 followed by a 7 days break.

In Part B of this trial, regorafenib will be administered continuously from Day 1 to Day 21. Only in Cycle 1, regorafenib dosing will start on Day 2 in order to assess the pharmacokinetics of pemetrexed and cisplatin without concomitant regorafenib dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Histological or cytological diagnosis of metastatic Stage IV or locally advanced, unresectable confirmed Stage IIIB nonsquamous Non-Small Cell Lung Cancer (NSCLC) not amenable to local therapy with curative intent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver, and renal function
* Controlled blood pressure [defined as systolic Blood Pressure (BP) <=150 mmHg and diastolic Blood Pressure (BP) <= 90 mmHg]
* Men and women of childbearing potential enrolled in this study must use adequate barrier birth control measures during the course of the study

Exclusion Criteria:

* Sensory neuropathy with sensory alterations or paresthesia (including tingling), interfering with function
* Hearing impairment
* Persistent proteinuria of Common Toxicity Criteria (CTC) Grade 3 or higher
* Cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II; patients must not have unstable angina (anginal symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months; cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Brain metastasis: patients with neurological symptoms should undergo a Computerized Tomography (CT) scan / Magnetic Resonance Imaging (MRI) of the brain to exclude any new or progressive brain metastasis. Patients with brain metastases are excluded from the trial
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication
* Pulmonary hemorrhage/bleeding event > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks prior to the start of study treatment. Clinically significant hemoptysis (1 teaspoon or more) in the past 3 months
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks prior to the start of study treatment
* Evidence or history of bleeding diathesis or coagulopathy
* Centrally located tumors with radiologic evidence (CT or MRI) of local invasion of major blood vessels
* The effect of third space fluid, such as pleural effusion and ascites, on pemetrexed is unknown. In patients with clinically significant third space fluid, consideration should be given to draining the effusion prior to study start
* Patients with phaeochromocytoma Excluded Therapies and Medications, Previous and Concomitant
* Prior treatment with a systemic chemotherapy for metastatic NSCLC. Patients who underwent prior systemic treatment or radiotherapy for NSCLC in a neoadjuvant or adjuvant setting are eligible, but no chemotherapy treatment within the last 6 month prior to study entry is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related toxicities and adverse events and change from baseline in vitals signs and laboratory parameters | 3 years (depending on the treatment duration of individual patients)
Pharmacokinetics assessments of Alimta, Cisplatin, and regorafenib in Cycle 1 and 2 | end of cycle 2

SECONDARY OUTCOMES:
Biomarkers (includes but not limited to plasma protein analysis of angiogenesis-related proteins, DNA mutational anaylsis of tumor tissue and plasma) | 3 years (depending on the treatment duration of individual patients)
Tumor Assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) every second cycle | 3 years (depending on the treatment duration of individual patients)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - New Haven, Connecticut
  - Las Vegas, Nevada
  - New York, New York
  - Chapel Hill, North Carolina

REFERENCES:
- [Derived] Hellmann MD, Sturm I, Trnkova ZJ, Lettieri J, Diefenbach K, Rizvi NA, Gettinger SN. Preliminary Safety, Pharmacokinetics, and Efficacy of Regorafenib, Cisplatin, and Pemetrexed in Patients With Advanced Nonsquamous Non-Small-Cell Lung Cancers. Clin Lung Cancer. 2015 Nov;16(6):514-22. doi: 10.1016/j.cllc.2015.04.003. Epub 2015 Apr 20. PMID 26003007